CLINICAL TRIAL: NCT05173129
Title: Comparison of Posture and Muscle Stiffness of Adolescent Boys With Haemophilia and Those of Age-matched Healthy Peers: a Controlled Cross-sectional Study
Brief Title: Posture Analysis for Patients With Haemophilia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Volkan Deniz, PT, Director, Cukurova University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 109/61
Record Dates: First submitted 2021-11-20; First posted 2021-12-29 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Hemophilia; Postural; Defect; Muscle Disorder
Keywords: haemophilia; posture; anti-gravity muscles; joint health
MeSH Terms: conditions — Hemophilia A; Muscular Diseases

STUDY DESIGN:
Intervention Model Description: cross-sectional study for two groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Haemophilic boys (Experimental): Adolescent boys with haemophilia
  Interventions: Diagnostic Test: Posture Analysis
- Healthy boys (Active Comparator): Healthy adolescent boys
  Interventions: Diagnostic Test: Posture Analysis

INTERVENTIONS:
Diagnostic Test: Posture Analysis — Posture analysis and assessment of mechanical properties of posture muscles

SUMMARY:
Hemophilia A and B are inherited disorders characterized by deficient or missing coagulation factors VIII or IX, respectively, of which the main long-term clinical manifestation is joint damage. Patients with haemophilia (PwH) are susceptible to clinical joint bleeding that may cause irreversible joint damage. Some degree of damage may already occur after the first haemarthrosis or even in children who never experienced clinically evident joint bleeds. Joints are mechanical systems with a structure strictly related to functioning. Therefore, any alteration in structure may have an impact on function (starting from the primary level of posture and anti-gravity muscles), which might in turn stress the joints and increase the risk of bleeding.The primary aim of this study is to investigate the changes in posture and the mechanical properties of anti-gravity muscles of adolescent PwH. The secondary aim is to determine the effect of joint dysfunction on posture in adolescent PwH.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent boys with haemophilia A or haemophilia B (for experimental group) and healthy adolescent boys (for control group).

Exclusion Criteria:

* To be with another congenital coagulopathy such as von Willebrand syndrome.
* To be unable to stand without support due to hemophilic arthropathy.
* To be having another musculoskeletal problem.
* To be having factor VIII or IX level in the plasma above 6%

Ages: 10 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Photogrammetry | Baseline
  The photogrammetry is a single evaluation method based on the analysis of two-dimensional photographs with a software.The erect-static posture of the participants will be analyzed with photogrammetry method. Firstly, two-dimensional photographs of the participant in the static-erect position will be taken.Afterwards, spinal and extremity angles will be measured in degrees using Kinovea™ software in the two-dimensional photographs transferred to the computer.
Myotonometric assessment | Baseline
  Myotonometric assessment is a reliable method in which the stiffness, elasticity and tone of the muscles are evaluated with a single measurement method.The mechanical properties (tone, stiffness, and elasticity) of the superficial muscles that affect posture will be evaluated with Myoton Pro™ device (Myoton AS, Tallinn, Estonia). With a single measurement made with Myoton Pro™ device, numerical values reflecting the mechanical properties of the muscle are obtained on the screen of the device.

SECONDARY OUTCOMES:
Haemophilia Joint Health Score | Baseline
  Joint health of adolescent patients with haemophilia will be assessed by Haemophilia Joint Health Score (HJHS). The HJHS, is calculated by adding the global gait score to the sum of 6 joint totals. The test could yield a minimum score of 0, which indicates healthy joint status, and a maximum score of 124 points (20 points per joint × 6+ 4 points for gait score), which indicates severe arthropathy in multiple joints

CONTACTS AND LOCATIONS:
Overall Officials: Nevin A Guzel, Prof. Dr., Study Director — Gazi University
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No